CLINICAL TRIAL: NCT01970735
Title: Clinical, Genetic and Epigenetic Characterization of Patients With FSHD Type 1 and FSHD Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-AOI-01
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FSHD patient (Experimental)
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test

SUMMARY:
The aim of the study was to compare the severity of illness between groups of patients (Facio-Scapulo-Humeral Dystrophy = FHSD1, FSHD2 and patients both FSHD1 and FSHD2).

Despite advances in research on the subject, answers are still needed on these diseases.

We also aim to determine whether the chromosomal genetic abnormality is involved in other diseases and the frequency of this mutation in the population of patients FSHD.

This study will increase our knowledge of the two forms of FSHD who present a common pathophysiological mechanism and may occur together in the same family with a worsening of the clinical phenotype worsening . In addition, epigenetic differences between FSHD type 1 and type 2 seems to have clinical consequences requiring appropriate management

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and <75 years
* FSHD patients 1 or 2 with or without genetic confirmation

Exclusion Criteria:

- Patient with all conditions considered by the investigator interfering with the proper conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2014-12-16 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
Muscle damage measure | One time at the inclusion
Level of muscle damage | One time at the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Archet 1, Nice, France

REFERENCES:
- [Derived] Sacconi S, Briand-Suleau A, Gros M, Baudoin C, Lemmers RJLF, Rondeau S, Lagha N, Nigumann P, Cambieri C, Puma A, Chapon F, Stojkovic T, Vial C, Bouhour F, Cao M, Pegoraro E, Petiot P, Behin A, Marc B, Eymard B, Echaniz-Laguna A, Laforet P, Salviati L, Jeanpierre M, Cristofari G, van der Maarel SM. FSHD1 and FSHD2 form a disease continuum. Neurology. 2019 May 7;92(19):e2273-e2285. doi: 10.1212/WNL.0000000000007456. Epub 2019 Apr 12. PMID 30979860